CLINICAL TRIAL: NCT05749835
Title: Effects of Thoracic Screw Manipulation in Patients With Cervical Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HAMZA REC/Letter- 01392
Record Dates: First submitted 2023-02-20; First posted 2023-03-01 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Cervical Radiculopathy
Keywords: pain; thoracic manipulation; sustained natural epiphyseal glides; neck disability index
MeSH Terms: conditions — Radiculopathy; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracic Manipulation and Sustained Natural Apophyseal Glides and conventional therapy (Experimental): After the segmental mobility examination of thoracic spine, the therapist will apply a high-velocity, end range screw thrust to a restricted segment of the thoracic spine as described by Maitland et al
  Interventions: Other: Thoracic Manipulation and Sustained Natural Apophyseal Glides and conventional therapy
- Sustained Natural Apophyseal Glides and conventional therapy (Experimental): Position of therapist: stands beside the patient, while his\her head is cradled between your body and your right forearm (when you stand at his\her right side). Gentle pressure is now applied in a ventral direction on the spinous process of C7 while the skull remains still due to the control of your right forearm. (The really gentle moving force to do this comes from your left arm via the thenar eminence over the little finger on the spine of C7).
  Interventions: Other: Sustained Natural Apophyseal Glides and conventional therapy

INTERVENTIONS:
Other: Thoracic Manipulation and Sustained Natural Apophyseal Glides and conventional therapy — After the segmental mobility examination of thoracic spine, the therapist will apply a high-velocity, end range screw thrust to a restricted segment of the thoracic spine as described by Maitland.
  Arms: Thoracic Manipulation and Sustained Natural Apophyseal Glides and conventional therapy
Other: Sustained Natural Apophyseal Glides and conventional therapy — Position of therapist: stands beside the patient, while his\her head is cradled between your body and your right forearm (when you stand at his\her right side). Gentle pressure is now applied in a ventral direction on the spinous process of C7 while the skull remains still due to the control of your right forearm. (The really gentle moving force to do this comes from your left arm via the thenar eminence over the little finger on the spine of C7).
  Arms: Sustained Natural Apophyseal Glides and conventional therapy

SUMMARY:
Cervical radiculopathy is a pain and/or sensorimotor deficit syndrome that is defined as being caused by compression of a cervical nerve root. The compression can occur as a result of disc herniation, Spondylosis, instability, trauma, or rarely, tumors.

Thoracic spine manipulation (TSM) is defined as a high-velocity/low amplitude movement or "thrust" directed at any segment of the thoracic spine. Recent research has shown that Thoracic Joint Manipulation directed to the thoracic spine provides a therapeutic benefit to patients with neck pain and has been suggested as an appropriate strategy to minimize the risks associated with manipulation of the cervical spine

DETAILED DESCRIPTION:
Patient presentations can range from complaints of pain, numbness, and/or tingling in the upper extremity to electrical type pains or even weakness. Disc herniation accounts for 20-25% of the cases of cervical radiculopathy. Most of the time cervical radiculopathy appears unilaterally; however it is possible for bilateral symptoms to be present if severe bony spurs are present at one level, impinging/irritating the nerve root on both sides. If peripheral radiation of pain, weakness, or pins and needle are present, the location of the pain will follow back to the concerned affected nerve root Manual techniques include positional release technique, muscle energy technique, myofascial release technique, Cyriax technique, Natural Apophyseal Glides and Sustained Natural Apophyseal Glides, manual pressure release, proprioceptive neuromuscular facilitation and ischemic compression.

Thoracic spine manipulation (TSM) is defined as a high-velocity/low amplitude movement or "thrust" directed at any segment of the thoracic spine. Recent research has shown that Thoracic Joint Manipulation directed to the thoracic spine provides a therapeutic benefit to patients with neck pain and has been suggested as an appropriate strategy to minimize the risks associated with manipulation of the cervical spine

ELIGIBILITY:
Inclusion Criteria:

* Patients complaint from pain in the cervical spine and pain or paresthesia traveling from the neck into a specific region of the arm, forearm or hand
* Cervical Lateral flexion and rotation <60 degree
* Positive scores on 3 of 4 clinical tests: Spurling's test, upper-limb neurodynamic test/median nerve bias, cervical distraction test, and cervical rotation toward the symptomatic side of less than 60°
* Hypomobility at T1- T5 thoracic vertebrae on springing test.

Exclusion Criteria:

* Participants with a history of vertebro-basilary artery insufficiency.
* Patient with history of cervical surgery or arthroplasty
* Patients with a positive history of trauma, fracture or surgery of the cervical
* spine
* Diagnosed cases of Torticollis, and scoliosis
* History of osteoporosis, Any heart disease

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
NPRS (Numeric Pain Rating Scale). | four weeks
  The Numeric Pain Rating Scale (NPRS) measures the subjective intensity of pain. The NPRS is an eleven-point scale from 0 to 10. "0" = no pain and "10" = the most intense pain imaginable.
Inclinometer | four weeks
  Inclinometers are portable, lightweight, and inexpensive pieces of equipment that are used to measure range of motion, like goniometry. Inclinometers are used as a part of a physical examination. An intraclass correlation coefficient (ICC) was found to be between 0.87-0.95.
(Neck Disability Index) Urdu | four weeks
  the neck disability index is a ten-item self-reported Questionnaire that assesses pain and associated disability, with a total max score of 50 points. An Urdu version of neck disability index will be used in this study. The total scores (ICC = 0.99) of the Neck Disability Index -Urdu.

CONTACTS AND LOCATIONS:
Overall Officials: maria Khalid, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- The Physiotherapy clinic Saidpur Road, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No